CLINICAL TRIAL: NCT05123027
Title: NIDA CTN-0107 Peer Intervention to Link Overdose Survivors to Treatment (PILOT)
Brief Title: Peer Intervention to Link Overdose Survivors to Treatment (PILOT)
Acronym: PILOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Drug Abuse Treatment Clinical Trials Network (Network); The Emmes Company, LLC (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kelly Barth, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00103441; 3UG1DA013727-20S5 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-11-17 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Opioid Overdose
Keywords: overdose; peer support
MeSH Terms: conditions — Opiate Overdose; Drug Overdose | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Intervention to Link Overdose Survivors to Treatment (PILOT) Peer (Experimental)
  Interventions: Behavioral: Peer Intervention to Link Overdose Survivors to Treatment (PILOT) Peer; Behavioral: Treatment As Usual Peer
- Treatment As Usual Peer (Active Comparator)
  Interventions: Behavioral: Treatment As Usual Peer

INTERVENTIONS:
Behavioral: Peer Intervention to Link Overdose Survivors to Treatment (PILOT) Peer — Participants will meet with the PILOT Peer consistently throughout the 6 months of study participation.
  Arms: Peer Intervention to Link Overdose Survivors to Treatment (PILOT) Peer
Behavioral: Treatment As Usual Peer — Participants will receive recovery resources and standard of care procedures specific to the Emergency Department.

SUMMARY:
The purpose of the Peer Intervention to Link Overdose Survivors to Treatment (PILOT) study is to improve outcomes for individuals after surviving an overdose involving opioids. This study will be comparing the enhanced peer intervention known as PILOT for overdose survivors with treatment as usual (TAU) provided in the Emergency Department.

ELIGIBILITY:
To be included in this study participants must:

1. Be 18 years of age or older at time of first contact by research staff (no upper age limit for inclusion).
2. Meet one of the following non-fatal overdose involving opioids (NFOO) criteria:

   1. Having presented to the Emergency Department for any health issue within the past 48 hours AND self-report having a known or suspected overdose involving opioids in the past 72 hours, OR
   2. Having presented to the Emergency Department within the past 48 hours for any SUD-related health issue, self-report having a known or suspected overdose involving opioids in the past 30 days
3. Be able to provide sufficient locator information, defined as identifying at least two individual contacts other than the participant.
4. Be able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study as determined by research staff.
5. Be willing and able to confirm future SUD treatment receipt as evidenced by 2 out of 3 of the following: (a) signing appropriate releases to for study staff to confirm treatment with follow-up provider; (b) having technology necessary to visualize medication bottles and transmit to study team utilizing HIPAA-compliant platform; and/or (c) able and willing to undergo toxicology tests (in person or via HIPAA-compliant videoconferencing).

Exclusion criteria include those who are:

1. Identified as having had an intentional overdose as the Index NFOO.
2. Actively suicidal at the time of screening (defined as current intention and/or plan for suicide attempt).
3. Unable to complete study baseline procedures due to medical or psychiatric condition.
4. Currently in jail, prison or in police custody at the time of the index ED visit or under current terms of civil commitment or guardianship (i.e., OHRP-defined prisoner status).
5. Previously randomized as a participant in this study - individuals may only be enrolled and randomized once.
6. Unwilling to follow study procedures (e.g., unable to provide sufficient locator information [defined as two contacts] or unavailable for follow-up assessments).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Barth, DO, Principal Investigator — Medical University of South Carolina
Locations (3):
- United States (3):
  - Mercy Health Youngstown, Youngstown, Ohio
  - Prisma Health Upstate, Greenville, South Carolina
  - Providence Regional Medical Center, Everett, Washington

IPD SHARING:
Plan to Share IPD: No
This study will comply with the NIH Data Sharing Policy and Implementation Guidance (https://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm) and the HEAL Public Access and Data Sharing Policy (https://www.nih.gov/research-training/medical-research-initiatives/heal-initiative/research/heal-public-access-data-sharing-policy).

REFERENCES:
- [Derived] Papa C, McClure EA, McCauley J, Haynes L, Matheson T, Jones R, Jennings L, Lawdahl T, Ward R, Brady K, Barth KS. Peer Intervention to Link Overdose Survivors to Treatment (PILOT): Protocol for a Multisite, Randomized Controlled Trial Conducted Within the National Institute on Drug Abuse Clinical Trials Network. JMIR Res Protoc. 2024 Sep 17;13:e60277. doi: 10.2196/60277. PMID 39288373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, controlled, parallel group design was implemented across three sites within the National Drug Abuse Treatment Clinical Trials Network (CTN): Prisma Health Systems (Southern Consortium Node); Mercy Health (Ohio Valley Node), and Providence Regional Medical Center (Pacific Northwest Node). From December 2021 through February 2024, 150 participants identified in the ED as opioid overdose survivors were approached to participate in the study.
Pre-assignment Details: Participants were identified and recruited from the ED at the time of ED admission (primary method of recruitment). Recruitment, approaching patients, screening, consent, and study procedures were completed in-person or remotely, utilizing HIPAA-compliant videoconferencing. Participants could be approached, screened and randomized after ED admission and could be randomized after screening had occurred in the ED.
Period: Overall Study
Arm/Group | Peer Intervention to Link Overdose Survivors to Treatment (PILOT) Peer | Treatment As Usual Peer
Started | 72 | 78
Completed | 48 | 50
Not Completed | 24 | 28
Not completed — Lost to Follow-up | 17 | 22
Not completed — Incarceration | 3 | 4
Not completed — Death | 2 | 2
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Intervention to Link Overdose Survivors to Treatment (PILOT) Peer | Treatment As Usual Peer | Total
Number analyzed (Participants) | 72 | 78 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 76 | 146
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (11.58) | 38.1 (11.28) | 38.7 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 30 | 51
  Male | 51 | 48 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 66 | 70 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 12 | 23
  White | 51 | 53 | 104
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 5 | 5 | 10
Baseline ORBC score [Mean (Standard Deviation); unit: units on a scale] | 12.6 (7.4) | 12 (7.9) | 12.3 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-reported Overdose Risk Behaviors at 180 Days (6 Months) After Index ED Admission
Description: Past month total score on the modified Overdose Risk Behavior Checklist (OBRC) at 180 days (6 months post-randomization) compared between experimental groups. The ORBC was a 13-item scale with 11 of the items used to generate a total score (ranging from 0-44); higher scores indicate greater frequency and number of overdose risk behaviors.
Time Frame: 180 days (6 months)
Population: Intent to treat analysis. All randomized subjects were included in the analysis. A participant contributed to the Day 180 estimate if they had all fixed effect covariates including baseline ORBC score and an ORBC score at Day 180
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PILOT Intervention Arm: In addition to usual care steps (TAU arm), also meets in the ED and over the next 180 days with PILOT peer with specialized training in overdose survivor engagement.
- Treatment as Usual (TAU) Arm: Receives routine clinical treatment in the ED including TAU peer support specialists able to provide Screening, Brief Intervention, Referral to Treatment (SBIRT) interventions for patients presenting with substance use disorders or substance-related issues.
Arm/Group | PILOT Intervention Arm | Treatment as Usual (TAU) Arm
Number analyzed (Participants) | 72 | 78
units on a scale | 4.5 (6.7) | 5.6 (7.8)
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) Arm; The primary outcome was analyzed with a longitudinal mixed effects negative binomial model incorporating the total score at earlier time points as well as 180 days. Fixed effect covariates included baseline score, treatment, days, site, stratum, and an interaction between treatment and days. A random effect was included to account for correlation within each participant; Test type: Superiority; p = 0.399, Mixed Models Analysis — Threshold for significance: p< 0.05; Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.30 to 1.62]

2. Secondary Outcome: Number of Steps Achieved Along a Modified SUD Cascade of Care
Description: Number of steps achieved along a modified substance use disorder (SUD) Cascade of Care (0-11 steps possible) at 180 days post-randomization (6 months). Higher scores are associated with better outcomes.
Time Frame: 180 days (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PILOT Intervention Arm | Treatment as Usual (TAU) Arm
Number analyzed (Participants) | 72 | 78
units on a scale | 4.4 (2.6) | 3.9 (2.5)
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) Arm; This was modeled similar to the primary outcome, an over dispersed Poisson regression model with fixed effect covariates for treatment arm, treatment days, site, and stratum with an interaction between treatment arm and treatment days. Note that no baseline score covariate was included as all participants will be considered to have achieved 0 steps at baseline. A random intercept was included for each subject to account for repeated measures; Test type: Superiority; p = 0.53, Mixed Models Analysis — Threshold for significance: p< 0.05; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.83 to 1.45]

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: Given the low-risk nature of this study, only select Adverse Events (AEs) and Serious Adverse Events (SAEs), collectively termed Safety Events were tracked and reported. Accordingly, Safety Events associated with participant death, post-index overdoses, ED visits, and hospitalizations were solicited during the 30-, 90-, 180-, and 210-day visits (or in-between visits if reported spontaneously). Reporting timeframes for Safety Events followed regulatory requirements.
Arm/Group | Peer Intervention to Link Overdose Survivors to Treatment (PILOT) Peer | Treatment As Usual Peer
All-Cause Mortality (participants affected / at risk) | 2/72 | 2/78
Serious Adverse Events (participants affected / at risk) | 21/72 | 18/78
Other Adverse Events (participants affected / at risk) | 0/72 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peer Intervention to Link Overdose Survivors to Treatment (PILOT) Peer (N=72) | Treatment As Usual Peer (N=78)
Death (General disorders) | 0 | 1 — Unknown cause of death
Death (Cardiac disorders) | 0 | 1 — Cardiac arrest
Death (Injury, poisoning and procedural complications) | 1 | 0 — Overdose
Death (General disorders) | 1 | 0 — Unknown cause of death
Hospitalization (Psychiatric disorders) | 0 | 1 — Altered Mental Status
Hospitalization (Injury, poisoning and procedural complications) | 0 | 1 — Overdose
Hospitalization (Psychiatric disorders) | 0 | 1 — Psychiatric Evaluation
Hospitalization (Injury, poisoning and procedural complications) | 0 | 1 — Cocaine abuse, Suicidal Ideation
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Chest pain
Hospitalization (Infections and infestations) | 0 | 1 — Pain from wound infection
Hospitalization (General disorders) | 0 | 1 — Cancer
Hospitalization (Social circumstances) | 0 | 1 — Neck pain; Motor vehicle collision
Hospitalization (Infections and infestations) | 0 | 1 — Osteomyelitis/Discitis
Hospitalization (Infections and infestations) | 0 | 1 — Subacute bacterial endocarditis; drug overdose
Hospitalization (Psychiatric disorders) | 0 | 1 — Hallucination
Hospitalization (Psychiatric disorders) | 0 | 1 — Psychosocial stressors
Hospitalization (Psychiatric disorders) | 0 | 1 — Anxiety
Hospitalization (General disorders) | 0 | 1 — Self care deficit
Hospitalization (General disorders) | 0 | 1 — Mid-sternal chest pain; opioid withdrawal
Hospitalization (Cardiac disorders) | 0 | 1 — Acute on chronic congestive hearth failure
Hospitalization (Surgical and medical procedures) | 1 | 0 — Scheduled hip surgery
Hospitalization (Infections and infestations) | 1 | 0 — Wound infection post-surgery
Hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Pregnancy complication in 3rd trimester
Hospitalization (Injury, poisoning and procedural complications) | 1 | 0 — Drug overdose
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Double pneumonia/respiratory issues
Hospitalization (Psychiatric disorders) | 1 | 0 — Suicidal ideation
Hospitalization (Injury, poisoning and procedural complications) | 1 | 0 — Excessive use of ecstasy
Hospitalization (Psychiatric disorders) | 1 | 0 — Mental health problem
Hospitalization (Injury, poisoning and procedural complications) | 1 | 0 — Polysubstance abuse
Hospitalization (Psychiatric disorders) | 1 | 0 — Acute psychosis
Hospitalization (General disorders) | 1 | 0 — COVID positive
Hospitalization (Surgical and medical procedures) | 1 | 0 — Scheduled surgery
Hospitalization (Injury, poisoning and procedural complications) | 1 | 0 — Acute CVA; Accidental fentanyl overdose
Hospitalization (Infections and infestations) | 1 | 0 — Cellulitis of hand, right
Hospitalization (Renal and urinary disorders) | 1 | 0 — Rhabdomyolysis; Renal failure
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Acute respiratory failure; Asthma
Hospitalization (Renal and urinary disorders) | 1 | 0 — Rhabdomyolysis; Acute kidney injury

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT05123027/Prot_002.pdf
  • Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT05123027/SAP_003.pdf
  • Informed Consent Form (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT05123027/ICF_001.pdf